CLINICAL TRIAL: NCT00098553
Title: Phase II Trial Of RAD-001 In Metastatic Malignant Melanoma
Brief Title: Everolimus in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0377; NCI-2012-02640 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000402871 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- everolimus (Experimental): Patients receive oral everolimus once daily for 8 weeks. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.
  Patients are followed every 2 months until disease progression and then every 4 months for up to 5 years after registration.
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as everolimus, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Everolimus may also stop the growth of melanoma by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well everolimus works in treating patients with stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the median time to disease progression in patients with stage IV malignant melanoma treated with everolimus.

Secondary

* Determine the median overall survival of patients treated with this drug.
* Determine the clinical benefit rates (i.e., stable disease, partial remission, and complete response rates) in patients treated with this drug.
* Determine the toxicity profile of this drug in these patients.
* Determine changes in serum vascular endothelial growth factor levels in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral everolimus once daily for 8 weeks. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months until disease progression and then every 4 months for up to 5 years after registration.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant melanoma for which no known standard or potentially curative therapy exists or has been proven to extend life expectancy

  * Stage IV disease
* Measurable disease

  * At least 1 lesion ≥ 20 mm by CT scan or MRI OR ≥ 10 mm by spiral CT scan
* No intracranial disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* No bleeding diathesis

Hepatic

* AST ≤ 3 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3 ULN
* INR ≤ 1.5

Renal

* Creatinine ≤ 1.5 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing to refrain from foods high in fat content
* No uncontrolled infection
* No immunosuppression from any cause (e.g., known HIV infection)
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer treated with local resection only
* No other severe condition that would preclude study participation or compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior immunotherapy or biologic therapy

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No prior sirolimus or its analogues for any indication
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent steroids

Radiotherapy

* More than 4 weeks since prior radiotherapy to head and neck area
* More than 4 weeks since prior radiosurgery
* No prior radiotherapy to > 30% of bone marrow
* No concurrent radiotherapy

Surgery

* Not specified

Other

* At least 1 week since prior and no concurrent CYP3A4 inducers
* No concurrent warfarin
* No concurrent cytotoxic agents
* No other concurrent experimental drugs
* No other concurrent immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-04; Primary Completion 2007-07 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with progression-free disease at 16 weeks | at 16 weeks

SECONDARY OUTCOMES:
Median overall survival | Up to 5 years
Tumor response rate for 2 consecutive evaluations at least 8 weeks apart | Up to 5 years
Toxicity as measured by CTCAE v. 3.0 | Up to 5 years
disease progression | at 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ravi D. Rao, MD, MBBS, Study Chair — Mayo Clinic; Harold E. Windschitl, MD — Coborn Cancer Center; William J. Maples, MD — Mayo Clinic; Michael K. Gornet, MD — Mayo Clinic; James N. Ingle, MD — Mayo Clinic; Edward T. Creagan, MD — Mayo Clinic; Judith S. Kaur, MD — Mayo Clinic; Barbara A. Pockaj, MD — Mayo Clinic Hospital; Evanthia Galanis, MD — Mayo Clinic; Charles L. Loprinzi, MD — Mayo Clinic; Henry C. Pitot, MD — Mayo Clinic; Lori A. Erickson, MD — Mayo Clinic; Val J. Lowe, MD — Mayo Clinic
Locations (94):
- United States (94):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Trinity Medical Center - East, Moline, Illinois
  - Moline, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Green Bay Oncology, Limited - Iron Mountain, Iron Mountain, Michigan
  - Alexandria, Minnesota
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Brainerd Medical Center, Brainerd, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Adult and Pediatric Urology, P.L.L.P., Sartell, Minnesota
  - Saint Francis Cancer Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin

REFERENCES:
- [Result] Rao RD, Allred JB, Windschitl HE, et al.: N0377: results of NCCTG phase II trial of the mTOR inhibitor RAD-001 in metastatic melanoma. [Abstract] J Clin Oncol 25 (Suppl 18): A-8530, 479s, 2007.
- [Result] Rao RD, Windschitl HE, Allred JB, et al.: Phase II trial of the mTOR inhibitor everolimus (RAD-001) in metastatic melanoma. [Abstract] J Clin Oncol 24 (Suppl 18): A-8043, 463s, 2006.
- [Derived] Vera Aguilera J, Rao RD, Allred JB, Suman VJ, Windschitl HE, Kaur JS, Maples WJ, Lowe VJ, Creagan ET, Erickson LA, Markovic S. Phase II Study of Everolimus in Metastatic Malignant Melanoma (NCCTG-N0377, Alliance). Oncologist. 2018 Aug;23(8):887-e94. doi: 10.1634/theoncologist.2018-0100. Epub 2018 Apr 17. PMID 29666297